CLINICAL TRIAL: NCT03312517
Title: A Phase IV 3-Way Double-blind, Randomized, Crossover Study to Compare the Awakening Threshold Effects (Responsivity) of Belsomra 10 mg and 20 mg to Placebo in Non-elderly Insomniacs
Brief Title: Study to Compare the Awakening Threshold Effects of Belsomra 10 mg and 20 mg to Placebo in Non-elderly Insomniacs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Christopher Drake, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MISP 57338
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Insomnia
Keywords: insomnia; belsomra; suvorexant
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — suvorexant

STUDY DESIGN:
Intervention Model Description: double-blind, randomized 3-way crossover design
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study is double blinded. Investigator, participant, or care provider will be blinded to watch drug the subject receives during each treatment week.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Suvorexant 10mg (Active Comparator): Subjects will receive belsomra 10mg before bedtime. In the middle of the night, subjects will be awakened to auditory awakening tones.
  Interventions: Drug: Suvorexant 10 mg
- Suvorexant 20mg (Active Comparator): Subjects will receive belsomra 20mg before bedtime. In the middle of the night, subjects will be awakened to auditory awakening tones.
  Interventions: Drug: Suvorexant 20 mg
- Placebo oral capsule (Sham Comparator): Subjects will receive placebo before bedtime. In the middle of the night, subjects will be awakened to auditory awakening tones.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Suvorexant 10 mg — Subject will receive suvorexant 10mg
  Other Names: belsomra 10mg
  Arms: Suvorexant 10mg
Drug: Suvorexant 20 mg — Subject will receive suvorexant 20mg
  Other Names: Belsomra 20mg
  Arms: Suvorexant 20mg
Drug: Placebo oral capsule — Subject will receive placebo.
  Other Names: placebo
  Arms: Placebo oral capsule

SUMMARY:
Phase IV 3-Way Double-blind, Randomized, Crossover Study to Compare the Awakening Threshold Effects (responsivity) of Belsomra 10 mg and 20 mg to Placebo in non-elderly Insomniacs

DETAILED DESCRIPTION:
The study is an interventional single site study using a double blind, randomized 3-way crossover design with Belsomra 10 mg and 20 mg compared to a placebo. The total number of enrolled patients proposed is 12. A cross-over design is utilized so participants will be exposed to all treatment conditions in a controlled order (Belsomra 10 mg, 20 mg and placebo). Both men and women with insomnia will be utilized as the study population to improve the generalizability of outcome data. Subjects with other sleep disorders or unstable medical/psychiatric disorders will be excluded from the trial. Inclusion criteria will be men and women >18 and < 65 years of age.

Subjects will be randomly assigned to treatment sequences using a Latin square design. After a subject has qualified for the study, the next sequentially available randomization number will be assigned. The subject will be administered study drug corresponding with this assigned number.

During the night of each respective Polysomnography (PSG) assessments, subjects will be awoken at the approximate T-max of the active drug (2.5 hrs), with a matching placebo condition at the same time point using an identical responsivity protocol for each condition. The rationale for this is that t-max represents the time of greatest potential risk for a hypnotic in terms of balance, responsivity, and memory. Responsivity will be assessed using the Auditory Awakening Threshold test (AAT) and will be measured at 2.5 hours post dose for the Belsomra 10 and 20 mg (BEL), and placebo (PBO) conditions. Responsivity will be assessed at the approximate time above immediately after 5 minutes of consolidated (without arousals) NREM ( Non- rapid eye movement) stage 2 sleep has occurred.

ELIGIBILITY:
Inclusion Criteria

* Meets DSM-5 ( Diagnostic and statistical manual) diagnostic criteria for insomnia disorder
* ISI ( Insomnia Severity Index) > 10
* Age >18 and < 65
* Negative audiological screening exam

Exclusion Criteria:

* BMI >35 kg/m2
* Have symptoms consistent with the diagnosis of any sleep disorder other than insomnia (e.g., sleep apnea, narcolepsy, periodic leg movements, or restless leg syndrome).
* Have a known or suspected diagnosis of Acquired Immune Deficiency Syndrome (AIDS), or have tested seropositive for human immunodeficiency virus (HIV) antibody or antigen previously.
* Have any clinically significant abnormal finding in physical examination, neurological assessment, vital signs, elevated body temperature, or clinical laboratory tests, as determined by the Investigator.
* Have a known or exaggerated pharmacological sensitivity, hypersensitivity, or intolerance to Belsomra.
* Currently taking CYP3A inhibitors.
* Positive breathalyzer test for alcohol at Screening, PSG Screening or any Treatment night, or a positive urine drug screen (for amphetamines, barbiturates, benzodiazepines, cocaine, opiates, or cannabinoids) at Screening;
* History of hearing difficulty (e.g., use of a hearing aid).
* Intends to use any medication including over-the-counter (OTC) medications that would interfere with normal sleep architecture (such as systemic steroids, beta-adrenergic blockers, amphetamines, modafinil, etc.);
* Self-reports use of products containing nicotine of greater than 15 cigarettes daily, or cannot avoid products containing nicotine during the normal sleep periods;
* Self report consumption of more than five alcoholic beverages on any one day or > 14 alcoholic beverages weekly over the past week;
* Have a history of epilepsy or serious head injury
* Average Time in Bed < 6.5 hrs.
* Have used prescribed or OTC medications within 7 days of screening (Day 0) or intend to use any prescription or OTC medication during the study that may interfere with the evaluation of the study drug. This restriction includes taking medications that affect the Central nervous system. Any chronic maintenance therapy should have been maintained at a stable dosing regimen for at least 30 days before screening and subjects must continue this regimen throughout the study.
* Have used an investigational drug within 30 days or five half lives (whichever is longer) before screening, or plans to use an investigational drug during the study or have used belsomra or zolpidem

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris L Drake, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Medical Center - Columbus, Novi, Michigan, United States

REFERENCES:
- [Background] Greenblatt DJ, Harmatz JS, Shader RI. Update on Psychotropic Drug Prescribing in the United States: 2014-2015. J Clin Psychopharmacol. 2018 Feb;38(1):1-4. doi: 10.1097/JCP.0000000000000831. No abstract available. PMID 29215384
- [Background] Bonnet MH, Webb WB, Barnard G. Effect of flurazepam, pentobarbital, and caffeine on arousal threshold. Sleep. 1979 Spring;1(3):271-9. doi: 10.1093/sleep/1.3.271. PMID 504872
- [Background] Johnson LC, Church MW, Seales DM, Rossiter VS. Auditory arousal thresholds of good sleepers and poor sleepers with and without flurazepam. Sleep. 1979 Spring;1(3):259-70. doi: 10.1093/sleep/1.3.259. PMID 228373
- [Background] Johnson LC, Spinweber CL, Webb SC, Muzet AG. Dose level effects of triazolam on sleep and response to a smoke detector alarm. Psychopharmacology (Berl). 1987;91(4):397-402. doi: 10.1007/BF00216003. PMID 3108921
- [Background] Drake CL, Durrence H, Cheng P, Roth T, Pillai V, Peterson EL, Singh M, Tran KM. Arousability and Fall Risk During Forced Awakenings From Nocturnal Sleep Among Healthy Males Following Administration of Zolpidem 10 mg and Doxepin 6 mg: A Randomized, Placebo-Controlled, Four-Way Crossover Trial. Sleep. 2017 Jul 1;40(7). doi: 10.1093/sleep/zsx086. PMID 28575467
- [Background] Bettica P, Squassante L, Zamuner S, Nucci G, Danker-Hopfe H, Ratti E. The orexin antagonist SB-649868 promotes and maintains sleep in men with primary insomnia. Sleep. 2012 Aug 1;35(8):1097-104. doi: 10.5665/sleep.1996. PMID 22851805
- [Background] Herring WJ, Snyder E, Budd K, Hutzelmann J, Snavely D, Liu K, Lines C, Roth T, Michelson D. Orexin receptor antagonism for treatment of insomnia: a randomized clinical trial of suvorexant. Neurology. 2012 Dec 4;79(23):2265-74. doi: 10.1212/WNL.0b013e31827688ee. Epub 2012 Nov 28. PMID 23197752
- [Background] Michelson D, Snyder E, Paradis E, Chengan-Liu M, Snavely DB, Hutzelmann J, Walsh JK, Krystal AD, Benca RM, Cohn M, Lines C, Roth T, Herring WJ. Safety and efficacy of suvorexant during 1-year treatment of insomnia with subsequent abrupt treatment discontinuation: a phase 3 randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2014 May;13(5):461-71. doi: 10.1016/S1474-4422(14)70053-5. Epub 2014 Mar 27. PMID 24680372
- [Background] Tannenbaum PL, Stevens J, Binns J, Savitz AT, Garson SL, Fox SV, Coleman P, Kuduk SD, Gotter AL, Marino M, Tye SJ, Uslaner JM, Winrow CJ, Renger JJ. Orexin receptor antagonist-induced sleep does not impair the ability to wake in response to emotionally salient acoustic stimuli in dogs. Front Behav Neurosci. 2014 May 16;8:182. doi: 10.3389/fnbeh.2014.00182. eCollection 2014. PMID 24904334
- [Background] Tannenbaum PL, Tye SJ, Stevens J, Gotter AL, Fox SV, Savitz AT, Coleman PJ, Uslaner JM, Kuduk SD, Hargreaves R, Winrow CJ, Renger JJ. Inhibition of Orexin Signaling Promotes Sleep Yet Preserves Salient Arousability in Monkeys. Sleep. 2016 Mar 1;39(3):603-12. doi: 10.5665/sleep.5536. PMID 26943466
- [Background] Manber R, Harvey A. Historical perspective and future directions in Cognitive Behavioral Therapy for insomnia and behavioral sleep medicine. Clin Psychol Rev. 2005 Jul;25(5):535-8. doi: 10.1016/j.cpr.2005.04.002. No abstract available. PMID 15950345
- [Background] Allen RP, Burchell BJ, MacDonald B, Hening WA, Earley CJ. Validation of the self-completed Cambridge-Hopkins questionnaire (CH-RLSq) for ascertainment of restless legs syndrome (RLS) in a population survey. Sleep Med. 2009 Dec;10(10):1097-100. doi: 10.1016/j.sleep.2008.10.007. Epub 2009 Feb 4. PMID 19195928
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Keefe FB, Johnson LC, Hunter EJ. EEG and autonomic response pattern during waking and sleep stages. Psychophysiology. 1971 Mar;8(2):198-212. doi: 10.1111/j.1469-8986.1971.tb00451.x. No abstract available. PMID 4326132
- [Background] Spinweber CL, Johnson LC. Effects of triazolam (0.5 mg) on sleep, performance, memory, and arousal threshold. Psychopharmacology (Berl). 1982;76(1):5-12. doi: 10.1007/BF00430746. PMID 6123129
- [Background] Bruck D, Thomas IR. Smoke alarms for sleeping adults who are hard-of-hearing: comparison of auditory, visual, and tactile signals. Ear Hear. 2009 Feb;30(1):73-80. doi: 10.1097/AUD.0b013e3181906f89. PMID 19125029
- [Background] Rosenthal L, Bishop C, Helmus T, Krstevska S, Roehrs T, Roth T. Auditory awakening thresholds in sleepy and alert individuals. Sleep. 1996 May;19(4):290-5. doi: 10.1093/sleep/19.4.290. PMID 8776786
- [Background] Busby KA, Mercier L, Pivik RT. Ontogenetic variations in auditory arousal threshold during sleep. Psychophysiology. 1994 Mar;31(2):182-8. doi: 10.1111/j.1469-8986.1994.tb01038.x. PMID 8153254
- [Derived] Drake CL, Kalmbach DA, Cheng P, Roth T, Tran KM, Cuamatzi-Castelan A, Atkinson R, Singh M, Tonnu CV, Fellman-Couture C. Can the Orexin Antagonist Suvorexant Preserve the Ability to Awaken to Auditory Stimuli While Improving Sleep? J Clin Sleep Med. 2019 Sep 15;15(9):1285-1291. doi: 10.5664/jcsm.7920. PMID 31538599

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Presence of insomnia determined by clinical interview performed by a physician board certified in sleep medicine
Groups:
- Placebo Then Suvorexant 10mg, Then Suvorexant 20mg: Subjects first received Placebo, then Suvorexant 10mg, then Suvorexant 20mg. Treatment was administered 30 min. before bedtime. In the middle of the night, subjects will be awakened to auditory awakening tones.
- Placebo, Then Suvorexant 20mg, Then Suvorexant 10mg: Subjects first received Placebo, then Suvorexant 20mg, then Suvorexant 10mg. Treatment was administered 30 min. before bedtime. In the middle of the night, subjects will be awakened to auditory awakening tones.
- Suvorexant 10, Then Placebo, Then Suvorexant 20: Subjects first received Suvorexant 10mg, then placebo, then Suvorexant 20mg. Treatment was administered 30 min. before bedtime. In the middle of the night, subjects will be awakened to auditory awakening tones.
- Suvorexant 10mg, Then Suvorexant 20mg, Then Placebo: Subjects first received Suvorexant 10mg, then Suvorexant 20mg, then placebo. Treatment was administered 30 min. before bedtime. In the middle of the night, subjects will be awakened to auditory awakening tones.
- Suvorexant 20mg, Placebo, Suvorexant 10mg: Subjects first received Suvorexant 20mg, placebo, then Suvorexant 10mg. Treatment was administered 30 min. before bedtime. In the middle of the night, subjects will be awakened to auditory awakening tones.
- Suvorexant 20, Suvorexant 10mg, Placebo: Subjects first received Suvorexant 20, then Suvorexant 10mg, then Placebo. Treatment was administered 30 min. before bedtime. In the middle of the night, subjects will be awakened to auditory awakening tones.
Period: Overall Study
Arm/Group | Placebo Then Suvorexant 10mg, Then Suvorexant 20mg | Placebo, Then Suvorexant 20mg, Then Suvorexant 10mg | Suvorexant 10, Then Placebo, Then Suvorexant 20 | Suvorexant 10mg, Then Suvorexant 20mg, Then Placebo | Suvorexant 20mg, Placebo, Suvorexant 10mg | Suvorexant 20, Suvorexant 10mg, Placebo
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Analyzed Sample: Crossover study, all subjects will receive belsomra 10mg, belsomra 20mg and placebo before bedtime in 3 separate overnights. In the middle of the night, subjects will be awakened to auditory awakening tones.
Arm/Group | Analyzed Sample
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Number of participants in analysis [Count of Participants; unit: Participants] | 12

OUTCOME MEASURES:

1. Primary Outcome: Auditory Awakening Threshold
Description: Subjects will be awakened during the night to auditory awakening tones.
Time Frame: 2.5 hours post-dose of each Study Drug administration
Population: We compared the odds of individuals sleeping through a 85-db stimulus in each condition. A generalized linear mixed model was used to estimate binary outcomes
Measure: Mean (Standard Deviation); unit: decibels (db)
Arm/Group | Suvorexant 10mg | Suvorexant 20mg | Placebo Oral Capsule
Number analyzed (Participants) | 12 | 12 | 12
decibels (db) | 74.17 (23.44) | 83.75 (20.24) | 79.17 (22.34)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Adverse Event were collected before and after every overnight. In addition, a Safety Follow-up 2 weeks after either study completion or study withdrawal was performed.
Groups:
- Placebo: All 12 subjects received placebo, 30 min before bedtime in one of the treatment nights. Order of treatment was assigned randomly. In the middle of the night, subjects were awakened to auditory awakening tones.
- Belsomra 20mg: All 12 subjects received belsomra 20mg, 30 min before bedtime in one of the treatment nights. Order of treatment was assigned randomly. In the middle of the night, subjects were awakened to auditory awakening tones.
- Belsomra 10mg: All 12 subjects received belsomra 10mg, 30 min before bedtime in one of the treatment nights. Order of treatment was assigned randomly. In the middle of the night, subjects were awakened to auditory awakening tones.
Arm/Group | Placebo | Belsomra 20mg | Belsomra 10mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Belsomra 20mg (N=12) | Belsomra 10mg (N=12)
Dry Mouth (Nervous system disorders) | NA | 1 (1) | NA
Anxiety (Psychiatric disorders) | NA | 1 (1) | NA
Upset (Psychiatric disorders) | NA | 1 (1) | NA
Dizziness (Nervous system disorders) | NA | 1 (1) | NA
Tingling sensation in arm (Nervous system disorders) | NA | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT03312517/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT03312517/SAP_001.pdf